CLINICAL TRIAL: NCT04095156
Title: PLA2R Autoreactive B-Cell Subsets and Immune Cell Monitoring in Membranous Nephropathy: Identification of Outcome Predictors and Novel Insights Into Disease Pathogenesis
Brief Title: Autoreactive B Cells in Membranous Nephropathy
Acronym: PEPTIDE
Status: Recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: PEPTIDE
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Membranous Nephropathy
Keywords: Membranous nephropathy; B cells; Anti-PLA2R; Anti-CD20 antibodies
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A research biobank will be established at "Centro di Risorse Biologiche Mario Negri - Biobanca Malattie Rare" containing biological material in the form serum and peripheral blood mononuclear cell (PBMC) samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prospective cohort: Patients with biopsy-proven idiopathic MN, who are candidate to receive a B-cell depleting treatment as per center clinical practice.
  Interventions: Diagnostic Test: In vitro assays.
- Retrospective cohort: Patients with biopsy-proven idiopathic MN, who already received a B-cell depleting treatment as per center clinical practice.
  Interventions: Diagnostic Test: In vitro assays.
- Healthy volunteers cohort: Subjects > 18 years not known to suffer of any significant illness, not assuming any medication or drug on a regular basis.
  Interventions: Diagnostic Test: In vitro assays.

INTERVENTIONS:
Diagnostic Test: In vitro assays. — Biochemical and flow-cytometry analysis of specimen collected.

SUMMARY:
Membranous nephropathy (MN) is the most frequent cause of nephrotic syndrome (NS) in adults. The majority of MN patients show detectable circulating antibodies against the M-type phospholipase A2 receptor (PLA2R). Infusion of anti-CD20 monoclonal antibodies results in a profound depletion of B-cells, which are thought to be responsible for anti-PLA2R production. B-cell depletion is followed by NS remission in 70% of cases. Limited evidence highlighted that differences in the B- and T-cell compartments may exist between responders and non-responders. Owing to the non-homogenous efficacy of anti-CD20 treatment, investigators hypothesize that in MN patients who experience NS remission after B-cell depleting therapy, autoreactive B-cells may be mostly circulating, whereas in patients who do not respond to the same treatment, autoreactive B-cells may chiefly reside into secondary lymphoid organs - and thus be more resistant to the drug action. Researchers will therefore extensively analyze the circulating immune repertoire of MN patients before and after the infusion of B-cell lineage depleting agents, assessing the presence of circulating PLA2R autoreactive B cells from appropriately stratified responder and non-responder patients. Patients and healthy controls will be enrolled in this study. Patients will be stratified according to gender, anti-PLA2R status, type of B-cell lineage depleting agent received and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients inclusion criteria

* Males and females.
* Adults (> 18 years old).
* Patients with biopsy-proven idiopathic MN, who are candidate to receive (prospective cohort) or who already received (retrospective cohort) a B-cell depleting treatment as per center clinical practice.
* Mental state is such that they are able to understand and give valid consent to the study;
* Written informed consent according to the guidelines of the Declaration of Helsinki.

Healthy volunteers inclusion criteria

* Male and female (>18 years) not known to suffer of any significant illness;
* Not assuming any medication or drug on a regular basis;
* Negative urine analysis (urine dipstick, multistick);
* Written informed consent according to the guidelines of the Declaration of Helsinki

Exclusion Criteria:

Patients exclusion criteria

* Reasonable possibility of a secondary cause of MN (e.g.systemic lupus erythematosus, active hepatitis B, malignancy, drugs such as gold salts and penicillamine).
* Legal incapacity, intellectual disability/mental retardation, dementia, uncooperative attitude or any other evidence that patient will not be able to understand the study procedures and aims and to give written informed consent.

Healthy volunteers exclusion criteria

- Legal incapacity, intellectual disability/mental retardation, dementia, uncooperative attitude or any other evidence that patient will not be able to understand the study procedures and aims and to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-proven idiopathic MN, who are candidate to receive (prospective cohort) or who already received (retrospective cohort) a B-cell depleting treatment as per center clinical practice and healthy volunteers as controls
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Differences between anti-PLA2R positive MN patients and anti-PLA2R negative MN patients and healthy controls in the frequency of anti-PLA2R autoreactive circulating B-cells. | Changes from baseline and 3,6,9,12 and 24 month.
Differences between anti-PLA2R positive MN patients and anti-PLA2R negative MN patients and healthy controls in the frequency of immunoglobulin- and cytokine-secreting circulating B-cell subsets in resting and stimulated conditions. | Changes from baseline and 3,6,9,12 and 24 month.
Differences between anti-PLA2R positive MN patients and anti-PLA2R negative MN patients and healthy controls in spontaneous / stimulated immunoglobulin (including anti-PLA2R) and cytokine release from circulating B-cell subpopulations. | Changes from baseline and 3,6,9,12 and 24 month.
Differences between MN patients and healthy controls, and between responders and non-responders in the frequency of circulating B-cell subpopulations. | Changes from baseline and 3,6,9,12 and 24 month.
Differences between MN patients and healthy controls, and between responders and non-responders in the frequency of circulating T-cell, NK-cell, monocyte and dendritic cell subpopulations. | Changes from baseline and 3,6,9,12 and 24 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare " Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: Undecided